CLINICAL TRIAL: NCT06597266
Title: Feasibility Study on Using Smart Templates, That Link Rectification Approaches to Particular Patient Characteristics, for Socket Fitting
Brief Title: Feasibility Study on Using Smart Templates, That Link Rectification Approaches to Particular Patient Characteristics, for Transtibial Prosthetic Socket Fitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Radii Devices Ltd (Unknown); Opcare Ltd (Unknown)
Responsible Party: Principal Investigator, Alex Dickinson, Professor of Biomechanical Engineering, University of Southampton
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRAS 313408 / HRA REC 22/YH/02; 10014827 (Other Grant/Funding Number: Innovate UK)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Transtibial Amputation; Prosthetic
Keywords: transtibial; CAD/CAM; design; prosthetic limb

STUDY DESIGN:
Intervention Model Description: Study using mixed quantitative/qualitative methodology of quantitative outcome assessment and qualitative semi-structured interviews. A slightly larger than usual number of participants is used based on a power calculation for preliminary assessment of a secondary outcome measure, Socket Comfort Score.
Who Masked: Participant
Masking Description: Prosthetic sockets compared between the two arms are visually identical except for the fine details of their shape (i.e. the design) and participants will not be informed which is which, at the point of assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (evidence-generated socket) then Active Comparator (control socket) (Experimental): Participants are first fitted with an evidence-generated prosthetic check socket (experimental), and then fitted with a prosthetist-led prosthetic check socket (active comparator)
  Interventions: Device: Smart template - designed prosthetic check socket; Device: Clinician-designed prosthetic check socket
- Active Comparator (control socket) then Experimental (evidence-generated socket) (Experimental): Participants are first fitted with a prosthetist-led prosthetic check socket (active comparator), and then fitted with an evidence-generated prosthetic check socket (experimental)
  Interventions: Device: Smart template - designed prosthetic check socket; Device: Clinician-designed prosthetic check socket

INTERVENTIONS:
Device: Smart template - designed prosthetic check socket — Evidence-generated trial prosthetic sockets are designed automatically by performing machine learning analysis of past socket designs that were produced by expert clinicians, the participant's residual limb size and shape descriptors and patient descriptors
Device: Clinician-designed prosthetic check socket — Active comparator prosthetic sockets are designed by expert prosthetists, bespoke to the participant, in a computer aided design environment (CAD)

SUMMARY:
Prosthetic socket comfort and fit is important in ensuring individuals with amputation can get the most use from their prosthetic limb. Researchers from the University of Southampton and a spin out company Radii Devices Ltd have been developing software based upon the cutting-edge of engineering design to support clinicians in the design of the socket.

The technology uses data from previous socket designs and limb shapes to develop and train the software, developed working with Opcare Ltd, a prosthetics provider. The software suggests appropriate socket design shapes (templates) that may be optimal based on previous designs and whether they have fit and been comfortable.

The aim of this study is to assess the feasibility of sockets designed by the Radii Devices software, and a preliminary comparison against socket designed by a clinician (known as a prosthetist). Combining qualitative (semi-structured interview) and quantitative (Socket Comfort) methods, will enable understanding of the strengths and limitations and inform further development of the Radii Devices technology into full design software for prosthetists that provides optimal socket design support.

This study is funded by an Innovate UK Biomedical Catalyst grant and will be carried out over a 6 month period at Oxford, Roehampton and Bristol Opcare NHS prosthetic services. Prosthetists at these services and patients with a below-knee amputation will be eligible to apply if they are interested. Participation will be split into two stages. In Stage One participants will be asked to trial two sockets (designed using different methods) at their fitting appointment instead of the usual one. If participants would like to participate in the second stage they will be asked about their experiences of socket fit and comfort in interviews, and within a short socket comfort diary for patients.

DETAILED DESCRIPTION:
A well-fitting, comfortable prosthetic socket is an urgent priority for the 170 million people worldwide with amputation as it stops people being able to achieve their goals and participate in society. For clinics providing sockets, there is an increasing demand for prosthetic limbs, increasing costs and a shortage of prosthetists (the people who fit the limbs to the patients). The prosthetic socket connects a person's remaining limb with the rest of the prosthetic limb. When a prosthetic socket does not fit properly, it causes skin irritation, blistering and in the worst cases, ulcers. It will also lead to patients avoiding prosthetic use altogether or repeat clinic visits. These sockets are complicated to design due to differences in patient limb shape, skin properties and ability to tolerate pressure. Therefore, there is a need to support prosthetists to achieve the best socket fit they can for the patient, quicker, and with fewer complications that can lead to patients not wanting to wear their prosthetic limb.

Socket design involves a process called rectification which aims to optimise comfort, stability and mobility for the prosthesis user. To achieve this, the prosthetist will remove material or add material to shape the final socket design. Rectification is a very complicated problem; yet there is currently little guidance or evidence to support the process. This leaves the socket dependent upon the skill and experience of the individual prosthetist, who require years of training and experience. Even then getting an optimal socket fit can take up to 9 clinic visits.

The development of evidence-based socket design to improve socket fit is a primary objective of the International Society for Prosthetics & Orthotics. Critical to this is the ability to use information about past socket designs to learn from and increase understanding of the socket design process. This need goes back many decades, with Klasson asking the following questions in 1982 which are still unsolved today:

* What is a good fit?
* What information is necessary to achieve a good fit?
* Which processing of the information is necessary to arrive at a good fit?

Since 2014, University of Southampton researchers have developed technology to meet the patient and clinic need, guided by input from prosthetics providers including Opcare, and patients. This work has so far resulted in world-leading research on analysing shape and optimising socket design and the spin out of a company (Radii Devices). As part of a collaboration with Opcare, in November 2019, a study was carried out to assess the current socket design software, understand current practice and how socket design could be supported. Five prosthetists of varying experience were recruited and key areas in which computer software can be improved were identified, including:

1. inclusion of more data to support design;
2. a more intuitive interface; and
3. the ability to adapt to individual clinician preferences.

Challenges include the complicated 3D shapes within socket design and how to get and visualise meaningful data about the design process. Researchers at the University of Southampton and Radii Devices have developed a process which uses computational geometry, data science and biomechanical engineering expertise to achieve this. The developed software learns from past socket designs to suggest optimal socket design for an individual patient. This software will be tested within this research study to compare it against Opcare's current design process. This will enable researchers to understand the strengths and weaknesses of the technology and inform the development of design software incorporating this technology in the best way to support socket design.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over
* Attend the Bristol, Oxford or Roehampton NHS Opcare prosthetic services
* Have had a transtibial amputation
* Deemed ready to cast for a new prosthesis by the clinical team as per usual care at the prosthetic centre
* Able to understand verbal and written English and provide informed consent

Exclusion Criteria:

* under the age of 18
* Have had an ankle disarticulation, Knee disarticulation or transfemoral amputation
* Contraindication to be fit for a prosthetic socket
* Unwilling to trial or unable to tolerate trialling two sockets at a fitting session
* Unable to answer verbal questions (as per normal fitting appointment) on their socket fitting and comfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview | 30 minutes beginning immediately after device provision (socket fitting session), and optionally again one month after the fitting session.
  To assess the feasibility of the smart templates device, by capturing participants' views and experiences of in-clinic fitting of two sockets designed in different ways, and general usability of their new prosthetic socket.
  The interview will be of approximately 30 minutes duration and administered immediately after the prosthetic socket fitting session (i.e. provision of the intervention) by the researcher, and optionally again one month later at a face-to-face meeting, telephone or video call

SECONDARY OUTCOMES:
Socket Comfort Score (SCS) | 30 minutes, i.e. at the end of the intervention provision (socket fitting session), and optionally daily over the subsequent one month
  To confirm the design and operating specifications of the smart templates device intervention, before beginning a full clinical trial, a self-reported survey related to prosthetic device comfort, on a 0-10 scale where 0 and 10 represented the most uncomfortable and the most comfortable socket imaginable, respectively.
  The SCS outcome measure is collected during the usual clinical pathway of prosthetic socket fitting session (i.e. at the time of provision of the intervention) by the researcher, which typically takes around 30 minutes. In this study it will be administered at fitting by the fitting-clinician, and the participant will be given the option to report it additionally daily, over the subsequent month, in a paper or electronic diary either posted back to the researchers, submitted on a webform or sent by WhatsApp.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dickinson, PhD, Principal Investigator — University of Southampton
Locations (3):
- United Kingdom (3):
  - Bristol Centre for Enablement, Bristol
  - Oxford Centre for Enablement, Oxford
  - Douglas Bader Rehabilitation Centre, Queen Mary's Hospital, Roehampton

IPD SHARING:
Plan to Share IPD: No
Requests for study data may be submitted to the University of Southampton's Research Governance Office once the results of the study have been published, and details for access requests will be included in the publication. Requests will be dealt with on a case by case basis and in accordance with the University of Southampton's standard procedures.

REFERENCES:
- [Background] A Comparison between Evidence-Generated Transtibial Sockets and Conventional CADCAM Designs, from the Patient's Perspective Florence Mbithi Dr, Maggie Donovan-Hall Prof, Jennifer Bramley Dr, Joshua Steer Dr, Charalambos Rossides Dr, Peter Worsley Prof, Chantel Ostler Dr, Cheryl Metcalf Prof, Dominic Hannett, Caroline Ward, Jack Kitchen, Sioned Steventon, Katy McIntosh, Shigong Guo Dr, Helen Harvey, David Henderson Slater Dr, Vijay Kolli Dr, Alex Dickinson Prof medRxiv 2024.09.17.24312762; doi: https://doi.org/10.1101/2024.09.17.24312762
- [Background] Dickinson AS, Steer JW, Rossides C, Diment LE, Mbithi FM, Bramley JL, Hannett D, Blinova J, Tankard Z, Worsley PR. Insights into the spectrum of transtibial prosthetic socket design from expert clinicians and their digital records. Front Rehabil Sci. 2024 Jul 12;5:1354069. doi: 10.3389/fresc.2024.1354069. eCollection 2024. PMID 39071770